CLINICAL TRIAL: NCT03229148
Title: Anesthesia Management in Endovascular Therapy for Ischemic Stroke: A Multicenter Randomised Study
Brief Title: Anesthesia Management in Endovascular Therapy for Ischemic Stroke
Acronym: AMETIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHU-343; 2017-0303001-90 (Other: 2017-0303001-90)
Record Dates: First submitted 2017-07-20; First posted 2017-07-25 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-07

CONDITIONS: Stroke; Thrombectomy; Anesthesia; Conscious Sedation
Keywords: Anesthesia or Conscious sedation for Thrombectomy for Stroke; Thrombectomy; Anesthesia; Conscious sedation; Stroke
MeSH Terms: conditions — Stroke | interventions — Anesthesia, General; Conscious Sedation

STUDY DESIGN:
Intervention Model Description: Multicentic, prospective, open, in parallel groups, stratified and randomised study.
Who Masked: Outcomes Assessor
Masking Description: It is an open label trial because it is not possible to maintain the anesthesiologist and patient blinded during the procedure. However, all subsequent evaluations will be conducted by clinical research staff blinded to the randomization group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anaesthesia (Active Comparator): In the general anesthesia group, rapid sequence induction is used. Conduction of general anesthesia and drugs used are left to the expertise of each investigating center. Systolic blood pressure has to be maintained between 140 and 180 mmHg with an intravenous norepinephrine infusion if necessary, tele-expiratory carbon dioxyde concentration (EtCO2) has to be maintained between 30 and 35 mmHg and SpO2 has to be maintained between 94 and 98 %.
  Interventions: Procedure: General anaesthesia
- Conscious Sedation (Active Comparator): In the conscious sedation group, drugs choice as well as pharmacological modulation will be left to the expertise of each investigating center. A sedation level between 0 and -3 with spontaneous breathing will be targeted, using the Richmond Agitation Sedation Scale (RASS) score validated in French. The lightest sedation level will be targeted, i.e. minimal to moderate sedation according to the US recommendations for sedation / analgesia. Systolic blood pressure will be maintained between 140 and 180 mmHg with an intravenous norepinephrine infusion if necessary and SpO2 will be maintained between 94 and 98%.
  Interventions: Procedure: Conscious Sedation

INTERVENTIONS:
Procedure: General anaesthesia — Procedure in which patients are induced into an unconscious state through use of various medications so that they do not feel pain during surgery
  Arms: General anaesthesia
Procedure: Conscious Sedation — A drug-induced depression of consciousness during which patients respond purposefully to verbal commands, either alone or accompanied by light tactile stimulation. No interventions are required to maintain a patent airway. (From: American Society of Anesthesiologists Practice Guidelines)
  Arms: Conscious Sedation

SUMMARY:
Objective of the study: to assess whether pharmacological sedation or general anesthesia for treatment of anterior circulation ischemic stroke with endovascular mechanical thrombectomy is associated with difference in morbidity (neurological outcome and peri-procedural complications).

DETAILED DESCRIPTION:
Since 2015, the management of anterior acute ischemic stroke (AIS) involves endovascular treatment with mechanical thrombectomy (MT). This urgent, difficult and uncomfortable procedure in frail patients requires multidisciplinary care ideally involving neurologists, interventional neuroradiologists and anesthesiologists.

Two anesthetic strategies are currently used: pharmacologic sedation in spontaneous ventilation or general anesthesia with tracheal intubation. General anesthesia provides strict immobility, protects the airway and avoids emergency intubation in case of severe procedural complication (notably vomiting and aspiration). Sedation is a frequently used alternative because of (1) a rapid execution which could reduce delay to reperfusion, (2) a lower risk of blood pressure drop that may compromise cerebral blood flow in the penumbra area, (3) the theoretical capacity to assess neurological status during the procedure and (4) the supposed risk of complications associated with mechanical ventilation and intravenous anesthestics on brain metabolism. Nevertheless, sedation exposes to dramatic complications in case of patient agitation and movements.

The choice of the ideal anesthesic management is still lacking. Old retrospective studies seemed to favor sedation with worst neurological outcome associated with general anesthesia. Nevertheless, these datas suffered methodological issues with selection bias: more severe patients based on NIHSS score were rather treated with general anesthesia and blood pressure was not controlled. Recent studies that demonstrated the benefit of MT did not include a specific anesthetic protocol and none of the studies currently available included a blood pressure management protocol that appears to be an essential component of cerebral perfusion. A subgroup analysis of the MR Clean study, including patients with an identical initial NIHSS score, did not find benefit from MT in patients with general anesthesia compared to those receiving sedation. Finally, authors concluded that performing a MT under general anesthesia would significantly lengthen the reperfusion delay and nullify the benefit of MT.

The prospective, randomized, single-center SIESTA trial, conducted in 150 patients with an anterior circulation AIS, found no difference in the early neurological improvement (primary endpoint), assessed on the change in NIHSS score between admission and the 24th hour, between the conscious sedation group and the general anesthesia group. There were a tendency for a better 3-month neurological outcome in the general anesthesia group (37% vs 18% of patients with a Modified Rankin score of 0-2 in the general anesthesia and conscious sedation groups respectively), but it was not possible to conclude due to a lack of statistical power.

Due to the increasing number of patients eligible for endovascular MT and the potential implication of these two anesthetic management on the functional outcome, a study comparing general anesthesia and sedation during a MT seems essential as specified in the recent updated American Stroke Association guidelines.

The objective of this study is to assess whether sedation or general anesthesia during endovascular treatment with mechanical thrombectomy is associated with a difference in morbidity (neurological outcome and peri-procedural complications), in anterior circulation AIS.

ELIGIBILITY:
Inclusion Criteria:

* Acute anterior circulation ischemic stroke (terminal portion of the internal carotid artery, middle cerebral artery), with indication for radiological mechanical thrombectomy assessed by the neurology / neuroradiology team
* Over 18 years of age
* Benefiting from an affiliation to the French Social Security system
* Patient or familly informed consent. In case of patient incapacity and no family present, and due to the emergency of the procedure, the patient may be included on the sole decision of the investigator (emergency procedure with subsequent differed consent).

Exclusion Criteria:

* Altered vigilance defined by score ≥ 2 at item 1a "level of consciousness" of the NIHSS score
* Altered previous autonomy, defined by a modified Rankin score (mRS)> 1
* Acute ischemic stroke of posterior circulation or anterior cerebral artery
* Associated brain haemorrhage
* Pregnant or nursing women
* Patient under law protection
* Stroke complicating another acute illness or postoperative stroke.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
composite of functional independence at 3 months and absence of medical complication occurring by day 7 after endovascular therapy for anterior circulation AIS | Day 90
  The primary outcome measure is a composite of functional independence at 3 months and absence of medical complication occurring by day 7 after endovascular therapy for anterior circulation AIS. Functional independence is defined as a mRS score 0 to 2 by day 90. Medical complications are defined as intervention-associated arterial perforation or dissection, pneumonia or myocardial infarction or acute cardiogenic pulmonary oedema or malignant stroke evolution occurring by day 7

SECONDARY OUTCOMES:
Ordinal score on the mRS by day 90 | at day 90
Functional independence by day 90 defined as a mRS score 0-2 | at day 90
Excellent recovery by day 90 defined as a mRS score 0-1 | at day 90
Moderate recovery by day 90 defined as a mRS score 0-3 | at day 90
Shift analysis of day 90 mRS adjusted for initial prognostic factors | at day 90
  (baseline mRS, age, initial NIHSS, carotid top occlusion)
Good recovery defined with sliding dichotomy responder analysis relating day 90 mRS with baseline NIHSS score: mRS 0 for NIHSS ≤ 7; mRS 0-1 for NIHSS 8-14; mRS 0-2 for NIHSS > 14 | at day 90
Intraprocedural hemodynamic and ventilatory conditions and complications defined as hypotension, blood pressure variability, hypoxemia and aspiration | at day 90
Intervention-associated vessel and others complications defined as arterial dissection or perforation, groin hematoma, embolization in another arterial territory | at day 90
Door to groin puncture delay | at day 90
Door to reperfusion delay | at day 90
Successful reperfusion defined by the modified Treatment In Cerebral Ischemia (mTICI) reperfusion scale of 2b or 3 (with a grade of 2b or 3 indicating reperfusion of > 50% of the affected territory) | at day 90
NIHSS by day 1 and day 7 | by day 1 and day 7
Stroke unit and hospital length of stay | at day 90
Medical complications by day 7 defined as pneumonia, acute cardiogenic pulmonary oedema, myocardial infarction, extra pulmonary infection, venous thromboembolism, new event of AIS, epilepsy, gastrointestinal bleeding or other symptomatic bleeding | at day 7
Malignant stroke evolution by day 7 | by day 7
Symptomatic intracranial haemorrhage by day 7 defined as brain haemorrhage on imaging associated with an increase of at least 4 points in the NIHSS score | by day 7
Unexpected intensive care unit admission by day 7 | by day 7
Mortality by day 7 and day 90 | by day 7 and day 90
Procedural feasibility score estimated by the radiologist and the anaesthesiologist and patient acceptability score | by day 7 and day 90

CONTACTS AND LOCATIONS:
Overall Officials: Russel Chabanne, MD, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne, France

REFERENCES:
- [Background] Berkhemer OA, Fransen PS, Beumer D, van den Berg LA, Lingsma HF, Yoo AJ, Schonewille WJ, Vos JA, Nederkoorn PJ, Wermer MJ, van Walderveen MA, Staals J, Hofmeijer J, van Oostayen JA, Lycklama a Nijeholt GJ, Boiten J, Brouwer PA, Emmer BJ, de Bruijn SF, van Dijk LC, Kappelle LJ, Lo RH, van Dijk EJ, de Vries J, de Kort PL, van Rooij WJ, van den Berg JS, van Hasselt BA, Aerden LA, Dallinga RJ, Visser MC, Bot JC, Vroomen PC, Eshghi O, Schreuder TH, Heijboer RJ, Keizer K, Tielbeek AV, den Hertog HM, Gerrits DG, van den Berg-Vos RM, Karas GB, Steyerberg EW, Flach HZ, Marquering HA, Sprengers ME, Jenniskens SF, Beenen LF, van den Berg R, Koudstaal PJ, van Zwam WH, Roos YB, van der Lugt A, van Oostenbrugge RJ, Majoie CB, Dippel DW; MR CLEAN Investigators. A randomized trial of intraarterial treatment for acute ischemic stroke. N Engl J Med. 2015 Jan 1;372(1):11-20. doi: 10.1056/NEJMoa1411587. Epub 2014 Dec 17. PMID 25517348
- [Background] Goyal M, Demchuk AM, Menon BK, Eesa M, Rempel JL, Thornton J, Roy D, Jovin TG, Willinsky RA, Sapkota BL, Dowlatshahi D, Frei DF, Kamal NR, Montanera WJ, Poppe AY, Ryckborst KJ, Silver FL, Shuaib A, Tampieri D, Williams D, Bang OY, Baxter BW, Burns PA, Choe H, Heo JH, Holmstedt CA, Jankowitz B, Kelly M, Linares G, Mandzia JL, Shankar J, Sohn SI, Swartz RH, Barber PA, Coutts SB, Smith EE, Morrish WF, Weill A, Subramaniam S, Mitha AP, Wong JH, Lowerison MW, Sajobi TT, Hill MD; ESCAPE Trial Investigators. Randomized assessment of rapid endovascular treatment of ischemic stroke. N Engl J Med. 2015 Mar 12;372(11):1019-30. doi: 10.1056/NEJMoa1414905. Epub 2015 Feb 11. PMID 25671798
- [Background] Saver JL, Goyal M, Bonafe A, Diener HC, Levy EI, Pereira VM, Albers GW, Cognard C, Cohen DJ, Hacke W, Jansen O, Jovin TG, Mattle HP, Nogueira RG, Siddiqui AH, Yavagal DR, Baxter BW, Devlin TG, Lopes DK, Reddy VK, du Mesnil de Rochemont R, Singer OC, Jahan R; SWIFT PRIME Investigators. Stent-retriever thrombectomy after intravenous t-PA vs. t-PA alone in stroke. N Engl J Med. 2015 Jun 11;372(24):2285-95. doi: 10.1056/NEJMoa1415061. Epub 2015 Apr 17. PMID 25882376
- [Background] Jovin TG, Chamorro A, Cobo E, de Miquel MA, Molina CA, Rovira A, San Roman L, Serena J, Abilleira S, Ribo M, Millan M, Urra X, Cardona P, Lopez-Cancio E, Tomasello A, Castano C, Blasco J, Aja L, Dorado L, Quesada H, Rubiera M, Hernandez-Perez M, Goyal M, Demchuk AM, von Kummer R, Gallofre M, Davalos A; REVASCAT Trial Investigators. Thrombectomy within 8 hours after symptom onset in ischemic stroke. N Engl J Med. 2015 Jun 11;372(24):2296-306. doi: 10.1056/NEJMoa1503780. Epub 2015 Apr 17. PMID 25882510
- [Background] Campbell BC, Mitchell PJ, Kleinig TJ, Dewey HM, Churilov L, Yassi N, Yan B, Dowling RJ, Parsons MW, Oxley TJ, Wu TY, Brooks M, Simpson MA, Miteff F, Levi CR, Krause M, Harrington TJ, Faulder KC, Steinfort BS, Priglinger M, Ang T, Scroop R, Barber PA, McGuinness B, Wijeratne T, Phan TG, Chong W, Chandra RV, Bladin CF, Badve M, Rice H, de Villiers L, Ma H, Desmond PM, Donnan GA, Davis SM; EXTEND-IA Investigators. Endovascular therapy for ischemic stroke with perfusion-imaging selection. N Engl J Med. 2015 Mar 12;372(11):1009-18. doi: 10.1056/NEJMoa1414792. Epub 2015 Feb 11. PMID 25671797
- [Background] Berkhemer OA, van den Berg LA, Fransen PS, Beumer D, Yoo AJ, Lingsma HF, Schonewille WJ, van den Berg R, Wermer MJ, Boiten J, Lycklama A Nijeholt GJ, Nederkoorn PJ, Hollmann MW, van Zwam WH, van der Lugt A, van Oostenbrugge RJ, Majoie CB, Dippel DW, Roos YB; MR CLEAN investigators. The effect of anesthetic management during intra-arterial therapy for acute stroke in MR CLEAN. Neurology. 2016 Aug 16;87(7):656-64. doi: 10.1212/WNL.0000000000002976. Epub 2016 Jul 15. PMID 27421546
- [Background] Schonenberger S, Uhlmann L, Hacke W, Schieber S, Mundiyanapurath S, Purrucker JC, Nagel S, Klose C, Pfaff J, Bendszus M, Ringleb PA, Kieser M, Mohlenbruch MA, Bosel J. Effect of Conscious Sedation vs General Anesthesia on Early Neurological Improvement Among Patients With Ischemic Stroke Undergoing Endovascular Thrombectomy: A Randomized Clinical Trial. JAMA. 2016 Nov 15;316(19):1986-1996. doi: 10.1001/jama.2016.16623. PMID 27785516
- [Background] Powers WJ, Derdeyn CP, Biller J, Coffey CS, Hoh BL, Jauch EC, Johnston KC, Johnston SC, Khalessi AA, Kidwell CS, Meschia JF, Ovbiagele B, Yavagal DR; American Heart Association Stroke Council. 2015 American Heart Association/American Stroke Association Focused Update of the 2013 Guidelines for the Early Management of Patients With Acute Ischemic Stroke Regarding Endovascular Treatment: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2015 Oct;46(10):3020-35. doi: 10.1161/STR.0000000000000074. Epub 2015 Jun 29. PMID 26123479
- [Derived] Chabanne R, Geeraerts T, Begard M, Balanca B, Rapido F, Degos V, Tavernier B, Molliex S, Velly L, Verdonk F, Lukaszewicz AC, Perrigault PF, Albucher JF, Cognard C, Guyot A, Fernandez C, Masgrau A, Moreno R, Ferrier A, Jaber S, Bazin JE, Pereira B, Futier E; ANARLF NetworkAMETIS Study Group. Outcomes After Endovascular Therapy With Procedural Sedation vs General Anesthesia in Patients With Acute Ischemic Stroke: The AMETIS Randomized Clinical Trial. JAMA Neurol. 2023 May 1;80(5):474-483. doi: 10.1001/jamaneurol.2023.0413. PMID 37010829
- [Derived] Tosello R, Riera R, Tosello G, Clezar CN, Amorim JE, Vasconcelos V, Joao BB, Flumignan RL. Type of anaesthesia for acute ischaemic stroke endovascular treatment. Cochrane Database Syst Rev. 2022 Jul 20;7(7):CD013690. doi: 10.1002/14651858.CD013690.pub2. PMID 35857365
- [Derived] Chabanne R, Begard M, Cazenave L, Pereira B. New paradigm shift in perioperative medicine: General anaesthesia finally better than procedural sedation for anterior circulation stroke thrombectomy? Anaesth Crit Care Pain Med. 2019 Dec;38(6):585-587. doi: 10.1016/j.accpm.2019.10.005. No abstract available. PMID 31785703
- [Derived] Chabanne R, Fernandez-Canal C, Degos V, Lukaszewicz AC, Velly L, Mrozek S, Perrigault PF, Molliex S, Tavernier B, Dahyot-Fizelier C, Verdonk F, Caumon E, Masgrau A, Begard M, Chabert E, Ferrier A, Jaber S, Bazin JE, Pereira B, Futier E; ANARLF Network and the AMETIS study group. Sedation versus general anaesthesia in endovascular therapy for anterior circulation acute ischaemic stroke: the multicentre randomised controlled AMETIS trial study protocol. BMJ Open. 2019 Sep 13;9(9):e027561. doi: 10.1136/bmjopen-2018-027561. PMID 31519668